CLINICAL TRIAL: NCT05759689
Title: The Effect of Fat Supplementation on the Appearance of Symptoms Associated With Dumping Syndrome in Patients Undergone Gastric Surgery
Brief Title: Fat Supplementation on Dumping Syndrome Related Symptoms After Gastric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, ATHANASIOS MIGDANIS, Research Associate Univeristy of Thessaly, Larissa University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LarissaUGH
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Dumping Syndrome; Gastric Surgery
Keywords: Dumping syndrome; Fat supplement; Gastric surgery
MeSH Terms: conditions — Dumping Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diagnose Dumping after supplement consumption (Experimental): Carbohydrate ingestion to provoke dumping syndrome related symptoms
  Interventions: Dietary Supplement: Dietary Supplement: Resource Energy; Dietary Supplement: Dietary Supplement: Calogen
- Fat supplementation (Active Comparator): A high fat supplement was added to the carbohydrate liquid meal that was previously used for diagnosis.
  Interventions: Dietary Supplement: Dietary Supplement: Resource Energy; Dietary Supplement: Dietary Supplement: Calogen

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Resource Energy — Carbohydrate Supplement
Dietary Supplement: Dietary Supplement: Calogen — Polyunsaturated liquid fat supplement

SUMMARY:
The purpose of the study is the investigation of the effect of fat supplement on gastric emptying rate and the appearance of symptoms of Dumping Syndrome in patients who have undergone gastrointestinal- duodenal surgery. Patients who have undergone bariatric surgery have been examined for the presence of the Dumping syndrome, with glucose measurements, the Sigstad's questionnaire and questionnaire of Arts. Patients diagnosed positive, reiterated the examination process in a second meeting consuming an extra fat supplement. The data obtained on the different appointments were compared between the two groups in a cross over design.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Dumping Syndrome

Exclusion Criteria:

* Patients with diabetes mellitus type 1 and 2
* Patients with impaired balance of fluids and electrolytes
* Patients on diuretics pills or corticosteroids or hypoglycemic tablets and Insulin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Glucose Levels | before the ingestion of the carbohydrate and fat supplement (baseline)
  Blood glucose measurement
Glucose Levels | 30 minutes after the ingestion of the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 60 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 90 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Glucose Levels | 120 minutes after the ingestion of the the carbohydrate and fat supplement
  Blood glucose measurement
Sigstad's Questionnaire | 1st hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Sigstad's Questionnaire | 2nd hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Arts's Questionnaire | 1st hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire
Arts's Questionnaire | 2nd hour after the ingestion of the supplements
  Dumping syndrome symptom associated questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Larissa, Larissa, Greece